CLINICAL TRIAL: NCT03979898
Title: Safety and Effectiveness of Autologous Adipose Tissue Derived Mesenchymal Stem Cell Implantation in Patients With Cerebral Palsy (CP)
Brief Title: Safety and Effectiveness of Autologous Adipose Tissue Derived Mesenchymal Stem Cell Implantation in Patients With CP
Acronym: CP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: R-Bio (Industry)
Collaborators: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: biostar-CP
Record Dates: First submitted 2016-08-01; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Astrostem (Experimental): Autologous Adipose Tissue Derived Mesenchymal Stem Cells
  Interventions: Biological: ASTROSTEM

INTERVENTIONS:
Biological: ASTROSTEM — Intravenous injection of Autologous Adipose derived mesenchymal stem cells. Dose : 15kg below : 0.5x10^7cells/5mL 15kg ~ 25kg : 1x10^8cells/10mL 25kg over : 1.5x10^8cells/15mL
  Other Names: Autologous Adipose Tissue Derived Mesenchymal Stem Cells

SUMMARY:
Safety and Effectiveness of Autologous Adipose Tissue Derived mesenchymal Stem Cell Implantation in Patients with CP

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of Adipose Tissue derived Mesenchymal stem cells (MSCs) in patient with Cerebral Palsy(CP)

ELIGIBILITY:
Inclusion Criteria:

* Children with spastic cerebral palsy of spastic paraplegia or quadriplegia involving the two side occurred at birth or before birth
* Age : 36 months - 12 year, males and females
* Subjects who understand and sign the consent form for this study
* Kaufman Assessment Battery for Children 50<K-ABC<100

Exclusion Criteria:

* The last three months had seizures or epilepsy patients taking the durg
* Genetic Diseases
* Recent cancer patients within 1 year
* patients witn a psychiatric disorder that may interfere in the clinical trial
* participating another clinical trials within 3 months
* Recently there is a change of the abrupt symptoms within three months of the patient
* Subjects with a infectious disease include HIV and VDRL
* Patients who penicillin hypersensitivity reactions
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria

Ages: 36 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Kaufman Assessment Battery for Children (K-ABC) | Baseline and 12 month
  Change from Baseline K-ABC at 12 months

SECONDARY OUTCOMES:
Blood concentration test | Baseline, 1, 3, 6 and 12 month
  Change from baseline concentration of dopamine, acetylcholine, serotonin at 1, 3, 6 and 12 month
Gross Motor Function Measurement (GMFM) | Baseline, 3, 6 and 12 month
  Change from Baseline GMFM at 12 months
Box and Block Test | Baseline, 3, 6 and 12 month
  Change from Baseline Box and block test at 12 months
Modified Ashworth Scale (MAS) | Baseline, 3, 6 and 12 month
  * Measurement of resistance during soft-tissue stretching
  * Scale range is 0(no increase in muscle ton) to 4(affected part rigid in flexion or extension)
  * Change from Baseline MAS at 12 months
SF-36 | Baseline, 3, 6 and 12 month
  * SF-36 is a survey to measure Mental & Physical Health
  * Score range is 0 to 100(the lower the score, the more disability)
  * Change from Baseline SF-36 at 12 months
Verification of ASTROSTEM's effect on the brain through fMRI & MRS (Magnetic Resonance Spectroscopy) scan | Baseline, 6 and 12 month
  Changes in fMRI & MRS scan from baseline to 6, 12 month
Kaufman Assessment Battery for Children (K-ABC) | Baseline and 6 month
  Change from Baseline K-ABC at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- KyungHee University Gandong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No